CLINICAL TRIAL: NCT05699980
Title: Prevalence and Comorbidities of Dermatoporosis: a French Prospective Observational Study in General Medicine Consultation
Status: Completed | Type: Observational
Sponsor: University of Lorraine (Other)
Collaborators: Study Director: Anne Claire Bursztejn, PHD-MD, CHU Nancy - University of Lorraine (Unknown); Study Chair: Christophe Goetz, MD, CHR Metz-Thionville - University of Lorraine (Unknown)
Responsible Party: Principal Investigator, Antoine Truchetet, Principal investigator, MD, University of Lorraine
Other Study IDs: University of Lorraine
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Dermatoporosis
Keywords: skin ageing; sun exposure; skin tears; purpura
MeSH Terms: conditions — Purpura

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient aged 60 or over presenting to their general practitioner: Patient aged 60 or over presenting to his general practitioner (among the 20 general practitioners recruited in Lorraine (eastern France))

SUMMARY:
The term dermatoporosis (DP) was proposed by JH. Saurat in 2004 and detailed in 2007 to describe a chronic cutaneous insufficiency and fragility syndrome.

The concept of DP, the positive diagnosis and the complications are well identified in the literature. However, while the consequences of skin aging are a growing concern, knowledge of DP is stagnant.

DP is clinically defined by the combination of three clinical signs: skin atrophy, white pseudo-scars, and senile purpura. It mainly sits on photo-exposed regions: posterior face of the forearms and back of the hands in 92 to 100% of cases; but also the pre-tibial, pre-sternal, and cephalic regions.

DP appears at around 60 years old and can worsen with advancing age. Complications of varying severity can occur during its development: skin tears, delayed healing, infection, hematomas including dissecting hematomas that are sometimes life-threatening.

DP is classified into four stages defined in 2004 and revised in 2012. The autonomy of the DP entity or its integration as a marker in multi-organ failure has not yet been determined. It is a condition on the borders of several specialties requiring good coordination between them (dermatologists, general practitioners, geriatricians, nurses, etc.)

The few published epidemiological studies report a prevalence ranging from 4% to 37.5% in patients aged 50 years and over. These epidemiological data are very heterogeneous (age of recruitment, patients hospitalized or seen on an outpatient basis in consultations of different specialties, sample of the population, etc.).

Among these studies, three clinical studies, two on a French hospital cohort, the other on outpatients in Dermatology in Finland, estimated the prevalence of DP between 27 and 32% in adults aged 60 years and older. In all three studies, DP was associated with advanced age, with a risk of DP up to double in patients aged 85 and older compared to younger patients. In two of these studies, a link was suggested with the status of chronic renal failure, either independently for one, or concomitant with taking anticoagulants and corticosteroids for the other. For Kluger et al., DP was also associated with the independent use of very strong local or systemic corticosteroids. For Chanca et al., an independent link between DP and tobacco consumption, taking anticoagulant treatment, and chronic recreational sun exposure has been observed.

DETAILED DESCRIPTION:
No clinical study has evaluated the prevalence of DP and the comorbidities often cited in adults aged 60 and over in general practice consultations.

The primary objective of this study is to assess the prevalence in a population aged 60 and over followed in a general practice in the North East of France (Lorraine). In addition, as it has been shown an association between DP and comorbidities or drug intake, the secondary objective is to investigate the possible existence of such associations.

Study design:

An observational, descriptive, transversal, multicenter study was conducted in the North East of France (Lorraine) between May and October 2022. We included by half-day, consecutively, all patients aged 60 and over presenting to a general medical consultation with 20 volunteer practitioners from the 4 Lorraine departments. Each practitioner was trained in the diagnosis of DP through a 27-minutes E-learning video and phone contacts.

Clinical and biological variables:

For each patient, the general practitioner performed his usual clinical examination, with a dermatological examination of the upper limbs. He completed an anonymous online questionnaire with data collected from the interrogation, medical files, and clinical examination.

The following data were reported: demographic data, active or former smoking, diabetes, dermatological history (atopic dermatitis, bullous dermatosis, psoriasis), chronic renal failure (MDRD < 60ml /min/m2), past sun exposure, Fitzpatrick phototype, treatments (anticoagulant, antiplatelet, systemic, local, inhaled corticosteroid therapy (cumulative duration >= 1 month)).

Finally, the signs of DP and the stage were filled in. For this study, we used the clinical staging of DP as proposed by Kaya and Saurat in 2012.

When signs of DP were present, photos of the dorsal aspect of the forearms and back of the hands (usual practice) were reviewed by the investigator and a dermatologist to confirm the diagnosis. The questionnaires were analyzed by the principal investigator.

As Chanca et al., we divided past sun exposure into three types: recreational, occupational, and childhood exposure. To assess chronic recreational sun exposure, patients were asked about past outdoor activities, such as walking or cycling at least 2 times/week. Occupational sun exposure was defined based on whether patients had an indoor or outdoor occupation. Childhood sun exposure was defined by a history of childhood sunburn.

Fitzpatrick phototype distinguishes six skin types based on tone, from very light skin that never tans (phototype 1), to dark skin, which never gets sunburn (phototype 6). According to this classification, we divided the patients into two categories: light skin (phototypes 1 to 3) and dark skin (phototypes 4 to 6).

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting to his general practitioner
* Patient aged 60 or over

Exclusion Criteria:

* Refusal of participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients aged 60 or over presenting to their general practitioner.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Presence or absence of dermatoporosis on the forearms or back of the hands | At admission, Day 1
  Presence or absence of dermatoporosis on the forearms or back of the hands in patients aged 60 or over in general practice

SECONDARY OUTCOMES:
Measurement of phototype | At admission, Day 1
  Measurement of phototype as a risk factor for dermatoporosis
Childhood sun exposure | At admission, Day 1
  Childhood sun exposure as a risk factor for dermatoporosis
Lifetime sun exposure Measurement of phototype | At admission, Day 1
  Lifetime sun exposure as a risk factor for dermatoporosis
Tobacco consumption | At admission, Day 1
  Tobacco consumption as a risk factor for dermatoporosis
Presence or absence of diabetes | At admission, Day 1
  Diabetes as a risk factor for dermatoporosis
Presence or absence of chronic renal failure | At admission, Day 1
  chronic renal failure as a risk factor for dermatoporosis
Presence or absence of antiplatelet consumption | At admission, Day 1
  antiplatelet consumption as a risk factor for dermatoporosis
Presence or absence of anticoagulant consumption | At admission, Day 1
  anticoagulant consumption as a risk factor for dermatoporosis
Presence or absence of systemic corticosteroid therapy | At admission, Day 1
  systemic corticosteroid therapy as a risk factor for dermatoporosis
Presence or absence of topical corticosteroid | At admission, Day 1
  topical corticosteroid on the forearms or back of the hands as a risk factor for dermatoporosis
Presence or absence of inhaled corticosteroid | At admission, Day 1
  inhaled corticosteroid as a risk factor for dermatoporosis

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Truchetet, MD, Principal Investigator — University of Lorraine; Anne Claire Bursztejn, PHD-MD, Study Director — CHU Nancy - University of Lorraine; Cédric Berbé, MD, Study Director — University of Lorraine; Christophe Goetz, MD, Study Chair — CHR Metz-Thionville - University of Lorraine
Locations (15):
- France (15):
  - Stéphanie Chevalier, Ancerville
  - Wissam Al Shouaib, Basse-Ham
  - Sophie LARUELLE, Bénaménil
  - Sophie Delaporte, Bulgnéville
  - Cédric Berbé, Cattenom
  - Sandra Pacini, Hayange
  - Anais Leclerc, Hettange-Grande
  - Benoit Nicolas, Hettange-Grande
  - Mathieu Zimmermann, Le Val-dAjol
  - Mélanie Damervalle, Longuyon
  - Patrick Vauthier, Longwy
  - Aurelie François, Raon-l'Étape
  - Jean-Louis Autissier, Thaon-les-Vosges
  - Cabinet Tronville en Barrois, Tronville-en-Barrois
  - Cabinet Varangéville, Varangéville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaya G, Saurat JH. Dermatoporosis: a chronic cutaneous insufficiency/fragility syndrome. Clinicopathological features, mechanisms, prevention and potential treatments. Dermatology. 2007;215(4):284-94. doi: 10.1159/000107621. PMID 17911985
- [Background] Mengeaud V, Dautezac-Vieu C, Josse G, Vellas B, Schmitt AM. Prevalence of dermatoporosis in elderly French hospital in-patients: a cross-sectional study. Br J Dermatol. 2012 Feb;166(2):442-3. doi: 10.1111/j.1365-2133.2011.10534.x. Epub 2011 Dec 5. No abstract available. PMID 21787367
- [Background] Chanca L, Fontaine J, Kerever S, Feneche Y, Forasassi C, Meaume S, Colboc H. Prevalence and risk factors of dermatoporosis in older adults in a rehabilitation hospital. J Am Geriatr Soc. 2022 Apr;70(4):1252-1256. doi: 10.1111/jgs.17618. Epub 2021 Dec 17. PMID 34918778
- [Background] Kluger N, Impivaara S. Prevalence of and risk factors for dermatoporosis: a prospective observational study of dermatology outpatients in a Finnish tertiary care hospital. J Eur Acad Dermatol Venereol. 2019 Feb;33(2):447-450. doi: 10.1111/jdv.15240. Epub 2018 Oct 1. PMID 30198583